CLINICAL TRIAL: NCT00699881
Title: Phase II Study of Cetuximab (Erbitux®) in Combination With Modified FOLFIRI in Patients With Advanced Gastric Cancer Who Failed to First-line Chemotherapy
Brief Title: Study of Cetuximab to Treat Gastric Cancer
Acronym: STAGE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Base for drug clinical trials, Fudan University cancer hospital, Department of medical oncology, Cancer Hospital, Fuandan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 62202- 806
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2008-06

CONDITIONS: Gastric Cancer
Keywords: Time to Progression; Toxicity; Overall survival; Response rate; Quality of live
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): administer cetuximab in combination with modified FOLFIRI
  Interventions: Drug: cetuximab

INTERVENTIONS:
Drug: cetuximab — cetuximab 400mg/m2 as initial dose, subsequently at 250mg/m2 weekly dose. CPT-11 180 mg/m2 CF 200 mg/m2 5Fu 400mg/m2 bolus, followed by 2.4g/m2 continuously intravenous infusion for 46 hours, days 1 and 15, every 4 weeks per cycle
  Other Names: treatment group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of cetuximab combined with FOLFIRI in patients with advanced gastric cancer who failed first-line chemotherapy

DETAILED DESCRIPTION:
Up to now, although FU based, cisplatin based and taxane based regimen, and ECF regimen have been suggested as the first line therapy for A/MGC by FDA, there is no standard regimen for patients with A/MGC as second line treatment. Based on the promising results of cetuximab combined with FOLFIRI in metastatic colorectal cancer, we design this clinical trial to evaluate the efficacy and safety of cetuximab combined with FOLFIRI for A/MGC patients as a second line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced or metastatic adenocarcinoma of the stomach
* ECOG performance scale ≤ 1
* At least one measurable lesion (larger than 10 mm in diameter by spiral CT scan)
* Adequate hepatic, renal, heart, and hematologic functions (platelets>80 × 109/L, neutrophil>2.0 × 109/L, serum creatinine ≤ 1.5mg/dl, total bilirubin within upper limit of normal(ULN), and serum transaminase≤2.5×the ULN)

Exclusion Criteria:

* Pregnant or lactating women
* Concurrent cancer
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Neuropathy, brain, or leptomeningeal involvement
* Uncontrolled significant comorbid conditions and previous radiotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
time to progression | every 8 weeks

SECONDARY OUTCOMES:
toxicity | every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, PhD, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Liu X, Guo W, Zhang W, Yin J, Zhang J, Zhu X, Liu T, Chen Z, Wang B, Chang J, Lv F, Hong X, Wang H, Wang J, Zhao X, Wu X, Li J. A multi-center phase II study and biomarker analysis of combined cetuximab and modified FOLFIRI as second-line treatment in patients with metastatic gastric cancer. BMC Cancer. 2017 Mar 14;17(1):188. doi: 10.1186/s12885-017-3174-z. PMID 28288572